CLINICAL TRIAL: NCT02129348
Title: Treatment of Psychosis and Agitation in Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Davangere P. Devanand, Professor of Clinical Psychiatry and Neurology, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: #6915; 1R01AG047146-01 (NIH)
Record Dates: First submitted 2014-04-29; First posted 2014-05-02 (Estimated); Results first posted 2021-08-16 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Alzheimer's Disease; Psychosis; Agitation
Keywords: Alzheimer's disease; psychosis; agitation; aggression; Lithium; delusions; hallucinations
MeSH Terms: conditions — Alzheimer Disease; Psychotic Disorders; Psychomotor Agitation; Aggression; Delusions; Hallucinations | interventions — Lithium; Lithium Carbonate

STUDY DESIGN:
Intervention Model Description: Participants were outpatients and recruited primarily from memory clinics and physician referrals at all four sites. Salient inclusion criteria were a diagnosis of possible or probable Alzheimer's disease by National Institute on Aging (NIA) criteria, score ≥4 on the Neuropsychiatric Inventory (NPI) domain score for agitation/aggression, Folstein Mini Mental State Exam (MMSE) range 5-26, and availability of an informant. Patients with current major depression or suicidality, alcohol/substance dependence in the prior 6 months, bipolar or other psychotic disorder, and specific neurological disorders were excluded.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients were randomized to lithium or placebo, 1:1, stratified by site, for 12 weeks. Randomization, developed by the statistician and executed by the NYSPI pharmacy, was stratified within each site by the presence of psychosis (NPI score ≥4 on delusions or hallucinations) with randomization sequences balanced in blocks of four.
  All study personnel and patients were masked to treatment assignment. After the final study visit, a psychiatrist independent of the study was unmasked and clinically treated the patient while study personnel remained blind.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lithium Treatment Group (Active Comparator): The patient will be started on lithium 150mg/day, with subsequent dose titration to 300mg/day at the 2-week visit, 450mg/day at the 4-week visit, and 600mg/day (maximum daily dose) if tolerated and based on lithium blood level. Blood will be drawn at each study visit. This upward dose titration will occur only if clinically indicated (absence of response at lower doses without intolerable side effects).
  Patients who develop side effects, e.g., tremor, falls, will have their dose reduced.
  Interventions: Drug: Lithium
- Placebo Group (Placebo Comparator): The patient will be started on placebo 150mg/day, with subsequent dose titration to 300mg/day at the 2-week visit, 450mg/day at the 4-week visit, and 600mg/day (maximum daily dose) if tolerated and based on sham lithium blood level. Blood will be drawn for sham lithium levels at weeks 2, 4, 6, 8, and 12. This upward dose titration will occur only if clinically indicated (absence of response at lower doses without intolerable side effects).
  Patients who develop side effects, e.g., tremor, falls, will have their dose reduced.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lithium
  Other Names: lithium carbonate
  Arms: Lithium Treatment Group
Drug: Placebo
  Arms: Placebo Group

SUMMARY:
Clinically, many patients with AD show no response or minimal response to antipsychotics for symptoms of agitation/aggression or psychosis, or they have intolerable side effects on these medications. Antipsychotics have a wide range of side effects, including the risk of increased mortality (60-70% higher rate of death on antipsychotic compared to placebo) that led to an FDA black box warning for patients with dementia; a more recent review and meta-analysis showed a 54% increased risk of mortality. In addition, some patients show only partial response to antipsychotics and symptoms persist. For these reasons, the investigators need to study alternative treatment strategies. Currently, there is no FDA-approved medication for the treatment of psychosis or agitation in AD.

The investigators innovative project will examine the efficacy and side effects of low dose lithium treatment of agitation/aggression with or without psychosis in 80 patients with AD in a randomized, doubleblind, placebo-controlled, 12-week trial (essentially a Phase II trial). The results will determine the potential for a large-scale clinical trial (Phase III) to establish the utility of lithium in these patients.

DETAILED DESCRIPTION:
Symptoms of psychosis or agitation are common in Alzheimer's disease. These symptoms are associated with distress for the patient, an increased burden for caregivers, more rapid cognitive decline, greater risk of institutionalization and mortality, and increased health care costs. In a recent meta-analysis, caregiver education and behavior modification studies revealed a small to medium effect size in treating agitation in these patients. However, none of these studies were double-blind (difficult to achieve in such studies) and none had a control group that received the same amount of staff time as the intervention group, thereby biasing the results toward the active intervention.

Among the psychotropic medications that have been studied, only antipsychotics have shown superiority over placebo for the treatment of psychosis and agitation in patients with dementia.

However, most studies show only moderate superiority for antipsychotic over placebo and a few studies have been negative. The side effects of antipsychotic medications include sedation, extrapyramidal signs, tardive dyskinesia, weight gain, and the metabolic syndrome. A pooled analysis from 17 short-term trials showed that the mortality rate in patients with dementia receiving antipsychotic medications was 1.6 to 1.7 times as high (60-70% increase in mortality rate) as the mortality rate in patients receiving placebo. These findings led the FDA to issue a black-box warning for antipsychotic medication use in patients with dementia; a more recent meta-analysis reported a slightly lower odds ratio of 1.54 (54% increase in mortality rate).

Lithium has several different actions from anticonvulsants, though both are effective in bipolar disorder, especially mania. Lithium is not being proposed here to treat mania in AD though the investigators will monitor symptoms on the Young Mania Rating Scale. In patients with AD, lithium has been studied for its putative cognitive enhancing effects. A few reports suggest that chronic lithium use reduces the risk of dementia, but other data show increased dementia risk with lithium use. A placebo-controlled, single-blind lithium trial showed no cognitive effects in patients with AD, but a recent trial of lithium in 45 patients with mild cognitive impairment (MCI, which often leads to clinically diagnosable AD) showed a small advantage for lithium (n=24) over placebo (n=21) in attention and other cognitive domains. None of these studies with lithium were intended to treat psychosis or agitation in AD, and patients with these symptoms typically were excluded in these clinical trials.

There has been no systematic placebo-controlled trial of lithium to treat agitation/aggression with or without psychosis in AD even though lithium is a highly effective treatment for mania with psychosis and symptoms of agitation or aggression. Nonetheless, the published studies of lithium to treat cognitive decline in older patients show that low-dose lithium is safe in patients with MCI or AD.

Specific Aims and Hypotheses Specific Aim 1. To compare changes in agitation/aggression with or without psychosis in patients with AD who receive 12 weeks of randomized, double-blind treatment with lithium or placebo.

Primary Hypothesis. Over these 12 weeks, the agitation/aggression domain score on the Neuropsychiatric Inventory (NPI) will decrease significantly more on lithium than placebo.

Secondary Hypothesis. Over these 12 weeks, the proportion of responders on lithium will be significantly greater than the proportion of responders on placebo. Response is defined as a 30% decrease in NPI core score (defined as the sum of domains for agitation/aggression, delusions and hallucinations) plus a CGI Change score of much improved or very much improved (CGI based on these behavioral symptoms only). Exploratory hypothesis. Over these 12 weeks, the psychosis score, measured by the sum of the NPI domain scores for delusions and hallucinations, will decrease significantly more on lithium than placebo. Specific Aim 2. To evaluate the tolerability of low dose lithium by assessing emergent somatic side effects over the course of the 12-week trial on lithium compared to placebo. Specific Aim 3. To explore associations between improvement on lithium (decrease in agitation/aggression and psychosis scores) and serum brain-derived neurotrophic factor (BDNF) levels (baseline, 12 weeks), a SNP in intron 1 of the ACCN1 gene, and variation at the 7q11.2 gene locus, because these indices are associated with lithium response in bipolar disorder. The investigators do not postulate a specific mechanism of action for lithium in the investigators trial, but will evaluate these three potential predictors of lithium response with the aim of improving patient selection for personalized treatment. The investigators will examine BDNF serum levels as a biomarker correlate of lithium treatment by correlating change in BDNF levels with change in NPI agitation/aggression and psychosis scores.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults.
2. Diagnosis of possible or probable AD by standard NIA criteria (McKahnn et al, 1984; McKhann et all, 2011)
3. Folstein MMSE 5-26 out of 30
4. Neuropsychiatric Inventory (NPI) agitation/aggression subscale score > 4. On each subscale (frequency X severity), a score higher than 4 represents moderate to severe symptoms.
5. Female patients need to be post-menopausal
6. Availability of informant; patients without an informant will not be recruited. Patients who lack capacity must have a surrogate.

Exclusion Criteria:

1. Medical contraindication to lithium treatment or prior history of intolerability to lithium treatment.

   Contraindications to lithium in this study include: resting tremor causing functional impairment, history of falls in the last month, untreated thyroid disease or any abnormal thyroid function test (T3, T4, or TSH), creatinine level greater than 1.5 mg/100ml or a glomerular filtration rate less than 44ml/min/ 1.73m2; blood pressure > 150/90 mm Hg; heart rate < 50 bpm; unstable cardiac disease based on history, physical examination, and ECG.
2. Medications, in combination with lithium, known to have adverse renal effects, including therapeutic or higher doses of diuretics, i.e. hydrochlorothiazide greater than 25mg daily or furosemide greater than 10mg daily. Whenever feasible, patients receiving concomitant antidepressants or antipsychotics will be washed off these medications for at least 24 hours before starting lithium. Patients who do not wish to discontinue antipsychotics or antidepressants, typically because of family member/caregiver objection, will be allowed to enter the trial provided there is no contraindication to concomitant lithium use with that specific psychotropic medication. During the trial, patients will be permitted to receive lorazepam as needed up to 1 mg/day for anxiety/insomnia, and non-benzodiazepine hypnotics, e.g., zolpidem.
3. Current clinical diagnosis of schizophrenia, schizoaffective disorder, other psychosis, or bipolar 1 disorder (DSM-IV TR criteria).
4. Current or recent (past 6 months) alcohol or substance dependence (DSM-IV TR criteria).
5. Current major depression or suicidality as assessed by the study psychiatrist.
6. Suicidal behavior or dangerous behavior with serious safety risk or risk of physical harm to self or others.
7. Parkinson's disease, Lewy body disease, multiple sclerosis, CNS infection, Huntington's disease, amyotrophic lateral sclerosis, other major neurological disorder.
8. Clinical stroke with residual neurological deficits. MRI findings of cerebrovascular disease (small infarcts, lacunes, periventricular disease) in the absence of clinical stroke with residual neurological deficits will not lead to exclusion.
9. Acute, severe, unstable medical illness. For cancer, patients with active illness or metastases will be excluded, but past history of successfully treated cancer will not lead to exclusion.
10. QTc interval > 460 ms at the time of baseline EKG is an exclusion criterion for treatment.
11. Hypernatremia as determined by serum sodium level > 150 meq/L.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2014-06; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: DP Devanand, MD, Principal Investigator — Columbia University
Locations (4):
- United States (4):
  - University of Miami Miller School of Medicine, Miami, Florida
  - McLean Hospital, Belmont, Massachusetts
  - New York State Psychiatric Institute, New York, New York
  - University of Texas Southwestern Medical Center, Dallas, Texas

REFERENCES:
- [Background] Devanand DP, Marder K, Michaels KS, Sackeim HA, Bell K, Sullivan MA, Cooper TB, Pelton GH, Mayeux R. A randomized, placebo-controlled dose-comparison trial of haloperidol for psychosis and disruptive behaviors in Alzheimer's disease. Am J Psychiatry. 1998 Nov;155(11):1512-20. doi: 10.1176/ajp.155.11.1512. PMID 9812111
- [Background] Camins A, Verdaguer E, Junyent F, Yeste-Velasco M, Pelegri C, Vilaplana J, Pallas M. Potential mechanisms involved in the prevention of neurodegenerative diseases by lithium. CNS Neurosci Ther. 2009 Winter;15(4):333-44. doi: 10.1111/j.1755-5949.2009.00086.x. PMID 19889130
- [Background] Devanand DP, Mintzer J, Schultz SK, Andrews HF, Sultzer DL, de la Pena D, Gupta S, Colon S, Schimming C, Pelton GH, Levin B. Relapse risk after discontinuation of risperidone in Alzheimer's disease. N Engl J Med. 2012 Oct 18;367(16):1497-507. doi: 10.1056/NEJMoa1114058. PMID 23075176
- [Background] Dunn N, Holmes C, Mullee M. Does lithium therapy protect against the onset of dementia? Alzheimer Dis Assoc Disord. 2005 Jan-Mar;19(1):20-2. doi: 10.1097/01.wad.0000155068.23937.9b. PMID 15764867
- [Background] Fahy S, Lawlor BA. Lithium use in octogenarians. Int J Geriatr Psychiatry. 2001 Oct;16(10):1000-3. doi: 10.1002/gps.452. PMID 11607946
- [Background] Forlenza OV, Diniz BS, Radanovic M, Santos FS, Talib LL, Gattaz WF. Disease-modifying properties of long-term lithium treatment for amnestic mild cognitive impairment: randomised controlled trial. Br J Psychiatry. 2011 May;198(5):351-6. doi: 10.1192/bjp.bp.110.080044. PMID 21525519
- [Background] Haddad P, Wieck A, Yarrow M, Denham P. 1999. The Lithium Side Effects Rating Scale (LISERS); development of a self-rating instrument. Eur Neuropsychopharmacol 9(s5): 231-232.
- [Background] Hampel H, Ewers M, Burger K, Annas P, Mortberg A, Bogstedt A, Frolich L, Schroder J, Schonknecht P, Riepe MW, Kraft I, Gasser T, Leyhe T, Moller HJ, Kurz A, Basun H. Lithium trial in Alzheimer's disease: a randomized, single-blind, placebo-controlled, multicenter 10-week study. J Clin Psychiatry. 2009 Jun;70(6):922-31. PMID 19573486
- [Background] Janowsky DS, Buneviciute J, Hu Q, Davis JM. Lithium-induced renal insufficiency: a longitudinal study of creatinine increases in intellectually disabled adults. J Clin Psychopharmacol. 2011 Dec;31(6):769-73. doi: 10.1097/JCP.0b013e31823607db. PMID 22020353
- [Background] Jefferson JW. A clinician's guide to monitoring kidney function in lithium-treated patients. J Clin Psychiatry. 2010 Sep;71(9):1153-7. doi: 10.4088/JCP.09m05917yel. PMID 20923621
- [Background] Katz I, de Deyn PP, Mintzer J, Greenspan A, Zhu Y, Brodaty H. The efficacy and safety of risperidone in the treatment of psychosis of Alzheimer's disease and mixed dementia: a meta-analysis of 4 placebo-controlled clinical trials. Int J Geriatr Psychiatry. 2007 May;22(5):475-84. doi: 10.1002/gps.1792. PMID 17471598
- [Background] Kessing LV, Sondergard L, Forman JL, Andersen PK. Lithium treatment and risk of dementia. Arch Gen Psychiatry. 2008 Nov;65(11):1331-5. doi: 10.1001/archpsyc.65.11.1331. PMID 18981345
- [Background] Macdonald A, Briggs K, Poppe M, Higgins A, Velayudhan L, Lovestone S. A feasibility and tolerability study of lithium in Alzheimer's disease. Int J Geriatr Psychiatry. 2008 Jul;23(7):704-11. doi: 10.1002/gps.1964. PMID 18181229
- [Background] McKnight RF, Adida M, Budge K, Stockton S, Goodwin GM, Geddes JR. Lithium toxicity profile: a systematic review and meta-analysis. Lancet. 2012 Feb 25;379(9817):721-8. doi: 10.1016/S0140-6736(11)61516-X. Epub 2012 Jan 20. PMID 22265699
- [Background] Nunes PV, Forlenza OV, Gattaz WF. Lithium and risk for Alzheimer's disease in elderly patients with bipolar disorder. Br J Psychiatry. 2007 Apr;190:359-60. doi: 10.1192/bjp.bp.106.029868. PMID 17401045
- [Background] Rej S, Abitbol R, Looper K, Segal M. Chronic renal failure in lithium-using geriatric patients: effects of lithium continuation versus discontinuation--a 60-month retrospective study. Int J Geriatr Psychiatry. 2013 May;28(5):450-3. doi: 10.1002/gps.3841. Epub 2012 Jun 4. PMID 22674617
- [Background] Schneider LS, Dagerman K, Insel PS. Efficacy and adverse effects of atypical antipsychotics for dementia: meta-analysis of randomized, placebo-controlled trials. Am J Geriatr Psychiatry. 2006 Mar;14(3):191-210. doi: 10.1097/01.JGP.0000200589.01396.6d. PMID 16505124
- [Background] Schneider LS, Dagerman KS, Insel P. Risk of death with atypical antipsychotic drug treatment for dementia: meta-analysis of randomized placebo-controlled trials. JAMA. 2005 Oct 19;294(15):1934-43. doi: 10.1001/jama.294.15.1934. PMID 16234500
- [Background] Shulman KI, Sykora K, Gill SS, Mamdani M, Anderson G, Marras C, Wodchis WP, Lee PE, Rochon P. New thyroxine treatment in older adults beginning lithium therapy: implications for clinical practice. Am J Geriatr Psychiatry. 2005 Apr;13(4):299-304. doi: 10.1176/appi.ajgp.13.4.299. PMID 15845755
- [Background] Tariot PN, Schneider LS, Cummings J, Thomas RG, Raman R, Jakimovich LJ, Loy R, Bartocci B, Fleisher A, Ismail MS, Porsteinsson A, Weiner M, Jack CR Jr, Thal L, Aisen PS; Alzheimer's Disease Cooperative Study Group. Chronic divalproex sodium to attenuate agitation and clinical progression of Alzheimer disease. Arch Gen Psychiatry. 2011 Aug;68(8):853-61. doi: 10.1001/archgenpsychiatry.2011.72. PMID 21810649
- [Background] Tredget J, Kirov A, Kirov G. Effects of chronic lithium treatment on renal function. J Affect Disord. 2010 Nov;126(3):436-40. doi: 10.1016/j.jad.2010.04.018. Epub 2010 May 16. PMID 20483164
- [Background] Wong YW, Tam S, So KF, Chen JY, Cheng WS, Luk KD, Tang SW, Young W. A three-month, open-label, single-arm trial evaluating the safety and pharmacokinetics of oral lithium in patients with chronic spinal cord injury. Spinal Cord. 2011 Jan;49(1):94-8. doi: 10.1038/sc.2010.69. Epub 2010 Jun 8. PMID 20531359
- [Background] Zhang X, Heng X, Li T, Li L, Yang D, Zhang X, Du Y, Doody RS, Le W. Long-term treatment with lithium alleviates memory deficits and reduces amyloid-beta production in an aged Alzheimer's disease transgenic mouse model. J Alzheimers Dis. 2011;24(4):739-49. doi: 10.3233/JAD-2011-101875. PMID 21321394
- [Derived] Deliyannides DA, Graff JA, Nino I, Lee S, Husain MM, Forester BP, Crocco E, Vahia IV, Devanand DP. Effects of lithium on serum Brain-Derived Neurotrophic Factor in Alzheimer's patients with agitation. Int J Geriatr Psychiatry. 2023 Sep;38(9):e6002. doi: 10.1002/gps.6002. PMID 37732619
- [Derived] Devanand DP, Crocco E, Forester BP, Husain MM, Lee S, Vahia IV, Andrews H, Simon-Pearson L, Imran N, Luca L, Huey ED, Deliyannides DA, Pelton GH. Low Dose Lithium Treatment of Behavioral Complications in Alzheimer's Disease: Lit-AD Randomized Clinical Trial. Am J Geriatr Psychiatry. 2022 Jan;30(1):32-42. doi: 10.1016/j.jagp.2021.04.014. Epub 2021 May 12. PMID 34059401
- [Derived] Devanand DP, Strickler JG, Huey ED, Crocco E, Forester BP, Husain MM, Vahia IV, Andrews H, Wall MM, Pelton GH. Lithium Treatment for Agitation in Alzheimer's disease (Lit-AD): Clinical rationale and study design. Contemp Clin Trials. 2018 Aug;71:33-39. doi: 10.1016/j.cct.2018.05.019. Epub 2018 May 31. PMID 29859917
- See also: Low Dose Lithium Treatment of Behavioral Complications in Alzheimer's Disease: Lit-AD Randomized Clinical Trial — https://pubmed.ncbi.nlm.nih.gov/34059401/

RESULTS

PARTICIPANT FLOW:
Groups:
- Lithium Treatment Group: The patient will be started on lithium 150mg/day, with subsequent dose titration to 300mg/day at the 2-week visit, 450mg/day at the 4-week visit, and 600mg/day (maximum daily dose) if tolerated and based on lithium blood level. Blood will be drawn at each study visit. This upward dose titration will occur only if clinically indicated (absence of response at lower doses without intolerable side effects).
  Patients who develop side effects, e.g., tremor, falls, will have their dose reduced.
  Lithium
- Placebo Group: The patient will be started on placebo 150mg/day, with subsequent dose titration to 300mg/day at the 2-week visit, 450mg/day at the 4-week visit, and 600mg/day (maximum daily dose) if tolerated and based on sham lithium blood level. Blood will be drawn for sham lithium levels at weeks 2, 4, 6, 8, and 12. This upward dose titration will occur only if clinically indicated (absence of response at lower doses without intolerable side effects).
  Patients who develop side effects, e.g., tremor, falls, will have their dose reduced.
  Placebo
Period: Overall Study
Arm/Group | Lithium Treatment Group | Placebo Group
Started | 38 | 39
Completed | 29 | 29
Not Completed | 9 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lithium Treatment Group | Placebo Group | Total
Number analyzed (Participants) | 38 | 39 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 34 | 36 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.6 (8.3) | 74.3 (6.9) | 74.9 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 46
  Male | 15 | 16 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 35 | 37 | 72
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 33 | 34 | 67
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 38 | 39 | 77
Neuropsychiatric Inventory (NPI) Agitation/Agression Domain [Mean (Standard Deviation); unit: units on a scale] — The primary outcome of Neuropsychiatric Inventory (NPI) Agitation/Aggression Domain was assessed at baseline, as were all secondary outcome measures.
  units on a scale | 7.7 (3.1) | 7.8 (2.9) | 7.75 (3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Neuropsychiatric Inventory (NPI) Agitation/Aggression Domain Score
Description: Neuropsychiatric Inventory (NPI) Agitation/Aggression Domain is the measure used that combines symptoms of agitation and aggression. Frequency X Severity rating score, range 0-12. Minimum score is 0, maximum score is 12. Higher score is a worse outcome and indicates more agitation and aggressive behavior.
Time Frame: Assessed at screening, Week 0, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Lithium Treatment Group | Placebo Group
Number analyzed (Participants) | 38 | 39
score on a scale | 3.2 [1.7 to 4.6] | 2.5 [1.1 to 4.0]
Statistical Analysis 1: Comparison: Lithium Treatment Group vs Placebo Group; Lithium will significantly reduce agitation/aggression compared to placebo. In intent-to-treat analyses, linear mixed effect models (MEM) were used to estimate means of change scores (baseline versus 12 weeks) by treatment group, lithium versus placebo, for continuous outcomes. The MEM method was used to incorporate all time-points of assessment and deal with missing data for participants who did not reach the 12-week time-point; Test type: Superiority; p = 0.53, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; Treatment Effect Difference = 0.7, 95% CI 2-sided [-1.4 to 2.7]

2. Secondary Outcome: Clinical Responder Defined as a 30% Decrease in NPI Core Score (Sum Score of NPI Domains of Agitation/Aggression, Delusions and Hallucinations) Together With a Clinical Global Impression (CGI) Behavior Change Score of 1 or 2
Description: The patient is classified as a responder (score=1) if both criteria are met or as a non-responder (score=0) if both criteria are not met. The first criterion to determine responder status, NPI core score, has a scoring range 0-36; each of the three component scores for symptoms of agitation/aggression, delusions and hallucinations has a scoring range 0-12. For each symptom and the total score, higher score indicates more symptoms. The second criterion to determine responder status, Clinical Global Impression (CGI), is used to assess change in overall behavior; scoring range 1-7 with higher scores indicating worsening over time and lower scores indicating improvement over time. Only patients who met both criteria, assessed as change compared to baseline, were counted as responders; all other patients were non-responders. Patients that demonstrated improvement at week 12 were reported; scores for earlier weeks were only used to assess progress throughout the study.
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Lithium Treatment Group | Placebo Group
Number analyzed (Participants) | 38 | 39
Participants | 12 | 7
Statistical Analysis 1: Comparison: Lithium Treatment Group vs Placebo Group; Change in both NPI core score (≥30% versus <30%) and CGI behavior change (1 or 2 versus ≥3) were required for response; these two measures were then analyzed separately. A x² test was used to identify whether there was a change in NPI core scores and CGI scores from baseline to week 12; Test type: Superiority; p = 0.26, Chi-squared — The threshold for statistical significance was p = 0.05; Treatment Effect Difference = 2.11, 95% CI 2-sided [0.73 to 6.13] — Odds ratio and its 95% confidence interval were computed

3. Secondary Outcome: Clinical Global Impression (CGI) Behavior Change
Description: Clinical Global Impression (CGI) Behavior Change score is the measure used to assess change in overall behavior; scoring range 1-7 with higher scores indicating worsening over time and lower scores indicating improvement over time. Scores ranging from 1-3 indicate improvement. Only patients that demonstrated improvement at week 12 were reported; scores for earlier weeks were only used to assess progress throughout the study.
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Lithium Treatment Group | Placebo Group
Number analyzed (Participants) | 38 | 39
Participants | 12 | 8
Statistical Analysis 1: Comparison: Lithium Treatment Group vs Placebo Group; CGI behavior change scores were categorized into responders versus non-responders (1 or 2 versus ≥3) using the last variable observation for drop-outs. A x² test was used to identify the percentage of participants in each group, lithium versus placebo, that improved from baseline to week 12; Test type: Superiority; p = 0.25, Chi-squared — The threshold of statistical significance was p = 0.05; Treatment Effect Difference = 1.79, 95% CI 2-sided [0.64 to 5.04]

4. Secondary Outcome: Young Mania Rating Scale
Description: Young Mania Rating Scale total score is the measure used to assess symptoms that occur in mania; each item is a symptom that is rated for severity. Scoring range 0-60. Minimum score is 0 and maximum score is 60. Higher scores mean a worse outcome.
Time Frame: Assessed at Week 0, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Lithium Treatment Group | Placebo Group
Number analyzed (Participants) | 38 | 39
score on a scale | 3.1 [0.9 to 5.3] | 1.1 [-1.1 to 3.3]
Statistical Analysis 1: Comparison: Lithium Treatment Group vs Placebo Group; In intent-to-treat analyses, linear mixed effect models (MEM) were used to estimate means of change scores (baseline versus 12 weeks) by treatment group, lithium versus placebo, for continuous outcomes. The MEM method was used to incorporate all time-points of assessment and deal with missing data for participants who did not reach the 12-week time-point; Test type: Superiority; p = 0.21, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; Treatment Effect Difference = 2.0, 95% CI 2-sided [-1.1 to 5.1]

5. Secondary Outcome: Treatment Emergent Signs and Symptoms
Description: Treatment Emergent Symptom Scale that covers 26 somatic symptoms, each rated as present (score=1) or absent (score=0). Total score is the measure used with scoring range 0-26; higher scores indicate more somatic symptoms.
Time Frame: Assessed at Week 0, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Lithium Treatment Group | Placebo Group
Number analyzed (Participants) | 38 | 39
score on a scale | 0.6 [-1.3 to 2.4] | 0.7 [-1.1 to 2.5]
Statistical Analysis 1: Comparison: Lithium Treatment Group vs Placebo Group; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.91, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; Treatment Effect Difference = -0.1, 95% CI 2-sided [-2.6 to 2.4]

6. Secondary Outcome: Simpson-Angus Scale
Description: Simpson Angus Scale for Extrapyramidal Sign requires in-person examination to assess gait, arm dropping, shoulder shaking, elbow rigidity, wrist rigidity, leg pendulousness, head dropping, glabella tap, tremor, and salivation. Total score is the measure used, range 0-40; higher scores indicate increased severity of signs.
Time Frame: Assessed at Week 0, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Lithium Treatment Group | Placebo Group
Number analyzed (Participants) | 38 | 39
score on a scale | -0.0 [-1.1 to 1.0] | 0.0 [-1.0 to 1.0]
Statistical Analysis 1: Comparison: Lithium Treatment Group vs Placebo Group; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.94, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; Treatment Effect Difference = 0.1, 95% CI 2-sided [-1.5 to 1.4] — Effect size (d)= -0.02 (Cohen's D)

7. Secondary Outcome: Basic Activities of Daily Living (BADL)
Description: Basic Activities of Daily Living with items for 6 functions: bathing, dressing, toileting, transferring, continence, and feeding. Each item is scored as unimpaired=1, impaired=0. Total score is the measure used, range 0-6; higher scores indicate better functioning.
Time Frame: Assessed at Week 0, Week2, Week 4, Week 6, Week 8, Week 10, Week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Lithium Treatment Group | Placebo Group
Number analyzed (Participants) | 38 | 39
score on a scale | 0.3 [-0.1 to 0.7] | 0.1 [-0.3 to 0.6]
Statistical Analysis 1: Comparison: Lithium Treatment Group vs Placebo Group; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.63, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; Treatment Effect Difference = 0.2, 95% CI 2-sided [-0.4 to 0.8]

8. Secondary Outcome: Zarit Caregiver Burden Interview
Description: Zarit Caregiver Burden Interview with the caregiver asked to rank 22 items on a scale with responses for each item from 'never' (score 0) to 'nearly always' (score 4). Total score is the measure used; range 0-88 with higher scores indicating greater caregiver burden.
Time Frame: Assessed at Week 0, Week 4, Week 8, Week 10, Week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Lithium Treatment Group | Placebo Group
Number analyzed (Participants) | 38 | 39
score on a scale | 2.8 [-1.1 to 6.6] | -0.4 [-4.2 to 3.3]
Statistical Analysis 1: Comparison: Lithium Treatment Group vs Placebo Group; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.24, Mixed Models Analysis — The threshold of statistical significance was p = 0.05; Treatment Effect Difference = 3.2, 95% CI 2-sided [-2.1 to 8.4] — Effect size (d)= 0.44 (Cohen's D)

9. Other Pre Specified Outcome: Folstein Mini-Mental Status Exam
Description: 30 item questionnaire used to assess degree of cognitive impairment. Orientation, registration, attention/calculation, recall, language, repetitions and commands are assessed. Total score is the measure used; range 0-30, higher scores indicate better global cognitive function.
Time Frame: Assessed at Screening, Week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Lithium Treatment Group | Placebo Group
Number analyzed (Participants) | 38 | 39
score on a scale | 0.9 [-0.3 to 2.2] | 0.9 [-0.4 to 2.1]
Statistical Analysis 1: Comparison: Lithium Treatment Group vs Placebo Group; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.96, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; Treatment Effect Difference = 0.0, 95% CI 2-sided [-1.7 to 1.8] — Cohen's d=0.01

10. Other Pre Specified Outcome: Severe Impairment Battery
Description: Neuropsychological test used to assess a patient's cognitive ability. The patient is asked to complete small tasks such as drawing shapes and printing their name. They are also asked to remember certain names and objects, such as a cup and a spoon, and the evaluator's first name. Total score is the measure used; range 0-100, higher scores indicate better cognition.
Time Frame: Assessed at Week 0, Week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Lithium Treatment Group | Placebo Group
Number analyzed (Participants) | 38 | 39
score on a scale | 2.1 [-1.1 to 5.4] | -0.0 [-3.3 to 3.2]
Statistical Analysis 1: Comparison: Lithium Treatment Group vs Placebo Group; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.35, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; Treatment Effect Difference = 2.2, 95% CI 2-sided [-2.3 to 6.6] — Cohen's d=0.35

ADVERSE EVENTS:
Time Frame: 12 weeks.
Description: Adverse events were based on self-report and caregiver report. Treatment Emergent Symptom Scale (TESS) total score was the measure for somatic side effects.
Arm/Group | Lithium Treatment Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/39
Serious Adverse Events (participants affected / at risk) | 11/38 | 11/39
Other Adverse Events (participants affected / at risk) | 30/38 | 33/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lithium Treatment Group (N=38) | Placebo Group (N=39)
Hypernatremia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Altered Mental Status (Psychiatric disorders) | 1 (1) | 0 (0)
Increased Agitation (Psychiatric disorders) | 3 (3) | 5 (5)
Fall (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypoglycemia (Endocrine disorders) | 1 (1) | 0 (0)
Dehydration (General disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Stomach Infection (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hyponatremia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Myoclonus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2.6% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lithium Treatment Group (N=38) | Placebo Group (N=39)
Increased Agitation (Psychiatric disorders) | 6 (6) | 11 (11)
Fall (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 4 (4)
Reduced Kidney Function (Renal and urinary disorders) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1)
Gait Instability (Nervous system disorders) | 4 (4) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 2 (2) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Tremor (Nervous system disorders) | 3 (3) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Contact Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Increased Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Increased Confusion (Psychiatric disorders) | 1 (1) | 1 (1)
Muscle Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Myoclonus (Nervous system disorders) | 1 (1) | 1 (1)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/48/NCT02129348/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/48/NCT02129348/SAP_001.pdf